CLINICAL TRIAL: NCT06759766
Title: Evaluation of Antimicrobial Potency of Garlic Lemon Extract Irrigant Versus Physiological Saline Irrigant Following Partial Pulpectomy in Primary Molars: A Randomized Clinical Trial
Brief Title: Evaluation of Antimicrobial Potency of Garlic Lemon Extract Irrigant Versus Physiological Saline Irrigant
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Yasser Yousef Mohamed, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU 30/12/2025
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Necrotic Primary Teeth

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial, parallel group, allocation ratio 1:1
Who Masked: Participant, Outcomes Assessor
Masking Description: The blinding of operator is not possible due to the nature of the material used. The clinical outcome assessor and statistician will be blinded in this study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Garlic-Lemon Extract irrigant (Active Comparator): garlic (Allium sativum) Shows a wide range of therapeutic effects due to the presence of allicin, ajoene & other thiosulfinates. It has antibacterial effect against wide range of gram-positive and gram-negative bacteria, anti-inflammatory, antioxidant, antiviral, antifungal, antitumor, immunomodulatory effects and tissue-dissolving capacity (Siddique, et al., 2020). According to (Elheeny., 2019) Allium sativum extract can be used efficiently as an irrigant for pulpectomy of primary molar root canals.
  Lemon (Citrus Limon) as well has curative properties such as, antibacterial, antiviral, antifungal, anti-inflammatory, anti-cancerous activities and removal of the smear layer as well. Due to presence of ascorbic acid, phenolic acids, polyphenols, and dietary fibers.
  the combination of Garlic-Lemon has been tested in adult teeth as an irrigant and showed an effective result equal to NaOCl (Siddique, et al., 2020).
  Interventions: Combination Product: Garlic-Lemon Extract irrigant
- physiological saline irrigant (Active Comparator): Normal saline solution exhibits no adverse effects on the developing successors; Serves primarily to facilitate root canal cleaning during the irrigation process, in comparison to other commercial synthetic irrigants such as Sodium hypochlorite (NaOCl), Chlorhexidine (CHX), Ethylenediamine tetra acetic acid (EDTA) which exhibit potential side effects and cytotoxic reactions (Sayadizadeh et al., 2019).
  Interventions: Other: physiological saline

INTERVENTIONS:
Combination Product: Garlic-Lemon Extract irrigant — garlic (Allium sativum) Shows a wide range of therapeutic effects due to the presence of allicin, ajoene & other thiosulfinates. It has antibacterial effect against wide range of gram-positive and gram-negative bacteria, anti-inflammatory, antioxidant, antiviral, antifungal, antitumor, immunomodulatory effects and tissue-dissolving capacity (Siddique, et al., 2020). According to (Elheeny., 2019) Allium sativum extract can be used efficiently as an irrigant for pulpectomy of primary molar root canals.
  Lemon (Citrus Limon) as well has curative properties such as, antibacterial, antiviral, antifungal, anti-inflammatory, anti-cancerous activities and removal of the smear layer as well. Due to presence of ascorbic acid, phenolic acids, polyphenols, and dietary fibers.
  the combination of Garlic-Lemon has been tested in adult teeth as an irrigant and showed an effective result equal to NaOCl (Siddique, et al., 2020).
  Arms: Garlic-Lemon Extract irrigant
Other: physiological saline — Normal saline solution exhibits no adverse effects on the developing successors; Serves primarily to facilitate root canal cleaning during the irrigation process, in comparison to other commercial synthetic irrigants such as Sodium hypochlorite (NaOCl), Chlorhexidine (CHX), Ethylenediamine tetra acetic acid (EDTA) which exhibit potential side effects and cytotoxic reactions (Sayadizadeh et al., 2019).
  Arms: physiological saline irrigant

SUMMARY:
To evaluate the antimicrobial potency of Garlic Lemon extract irrigant versus physiological saline irrigant following partial pulpectomy in primary molars.

DETAILED DESCRIPTION:
Pulpectomy is a suitable treatment of primary teeth with irreversible pulpitis, necrosis, or periodontitis due to caries or trauma. Due to the complex nature of the deciduous root canal system makes total removal of necrotic tissue by instrumentation alone impossible. Therefore, irrigation is a replenishing step to create a disinfectant atmosphere inside the root canal.

A variety of antiseptic and antibacterial irrigating solutions have been used such as (NaOCl), (CHX), and (EDTA). Due to their adverse effects, safety issues and cytotoxic reactions, Herbal products can be an alternative to these irrigants based on their previous history in medical field.

Herbal extracts such as garlic (Allium sativum) Shows a wide range of therapeutic effects due to the presence of allicin, ajoene & other thiosulfinates. It has antibacterial effect against wide range of gram-positive and gram-negative bacteria, anti-inflammatory, antioxidant, antiviral, antifungal, antitumor, immunomodulatory effects and tissue-dissolving capacity (Siddique, et al., 2020). According to (Elheeny., 2019) Allium sativum extract can be used efficiently as an irrigant for pulpectomy of primary molar root canals.

Lemon (Citrus Limon) as well has curative properties such as, antibacterial, antiviral, antifungal, anti-inflammatory, anti-cancerous activities and removal of the smear layer as well. Due to presence of ascorbic acid, phenolic acids, polyphenols, and dietary fibers.

the combination of Garlic-Lemon has been tested in adult teeth as an irrigant and showed an effective result equal to NaOCl (Siddique, et al., 2020).However, there is no studies have been performed to assess the combination of Garlic-lemon extract as an irrigant in deciduous molars.

ELIGIBILITY:
Inclusion Criteria:

1. The children's age range from four to seven years from both sexes.
2. Presence of localized swelling, sinus and pain on percussion which indicate non vital pulp.
3. Presence of periapical and furcation radiolucency in periapical radiograph.
4. Absence of history of systemic disease which would contraindicate pulp therapy e.g. infective endocarditis.
5. No previous history of antibiotics administration or last dose was taken from at least two weeks.

Exclusion Criteria:

1. Presence of advanced physiologic or pathologic root resorption in X-ray.
2. Uncooperative children.
3. Teeth with unrestorable crowns.
4. Teeth with abnormal anatomy and calcified canals.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
bacterial count | pre and after irrigation within the same visit
  colony forming unit (CFU) quantitative measure

CONTACTS AND LOCATIONS:
Overall Officials: Rasha M Hatem, Associate Professor, Study Director — Pediatric Department, Faculty of Dentistry, Cairo University.; Samaa S Hanafy, Lecturer, Study Director — Pediatric Department, Faculty of Dentistry, Cairo University.

REFERENCES:
- [Background] Elheeny AAH. Allium sativum extract as an irrigant in pulpectomy of primary molars: A 12-month short-term evaluation. Clin Exp Dent Res. 2019 Jun 26;5(4):420-426. doi: 10.1002/cre2.197. eCollection 2019 Aug. PMID 31452953
- [Background] Salem, M. R., Taha, S., & Abd El Gwad, R. (2017). Evaluation Of Antimicrobial Efficacy Of Green Tea Extract Irrigant Versus Physiological Saline Following Root Canal Treatment Of Infected Primary Molars In A Group Of Egyptian Children: A Randomized Clinical Trial. Egyptian Dental Journal, 63(Issue 1 - January (Orthodontics, Pediatric & Preventive Dentistry)), 101-110.
- [Background] Shalan, H. M. (2023). Evaluation of Antimicrobial Efficiency of Herbal Irrigants of Pulpectomized Primary Teeth. Mansoura Journal of Dentistry, 10(2), 97-101.
- [Background] Siddique, R., Anjaneyulu, K., & Muralidharan, N. P. (2019). Antimicrobial efficacy of garlic-lemon in comparison with sodium hypochlorite against E. faecalis. J Clin Diagn Res, 13(1), 55-58.
- [Background] Siddique R, Ranjan M, Jose J, Srivastav A, Rajakeerthi R, Kamath A. Clinical Quantitative Antibacterial Potency of Garlic-Lemon Against Sodium Hypochlorite in Infected Root Canals: A Double-blinded, Randomized, Controlled Clinical Trial. J Int Soc Prev Community Dent. 2020 Nov 24;10(6):771-778. doi: 10.4103/jispcd.JISPCD_287_20. eCollection 2020 Nov-Dec. PMID 33437712
- [Background] Sayadizadeh M, Shojaeipour R, Aminzadeh M, Horri A. Compare of the Combination of Saline and Chlorhexidine with Saline as Root Canal Irrigant in Pulpectomy of Primary Molars in 6-9 Years Old Children, A Double Blind Clinical Trial. J Dent Mater Tech 2019; 8(4): 174-181.
- [Background] Susila AV, Sai S, Sharma N, Balasubramaniam A, Veronica AK, Nivedhitha S. Can natural irrigants replace sodium hypochlorite? A systematic review. Clin Oral Investig. 2023 May;27(5):1831-1849. doi: 10.1007/s00784-023-04913-7. Epub 2023 Feb 18. PMID 36808559